CLINICAL TRIAL: NCT06224608
Title: Phase I Clinical Trial to Evaluate the Safety and Tolerability of Recombinant Mycobacterium Tuberculosis Fusion Protein (EEC) in Healthy Adults Aged 18-65 and Patients With Pulmonary Tuberculosis
Brief Title: Phase I Clinical Trial to Evaluate the Safety of Recombinant Mycobacterium Tuberculosis Fusion Protein (EEC) in Healthy Adults Aged 18-65 and Patients With Pulmonary Tuberculosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu CoenBiotech Co., Ltd (Industry)
Collaborators: Beijing Chest Hospital, Capital Medical University (Other); Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KN-EEC-I
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Tuberculosis
Keywords: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary tuberculosis patients (Experimental): Experimental drug of low-dose (2.5 μg/ml), medium-dose (5 μg/ml), and high-dose (10 μg/ml) will be conducted separately for 30 Pulmonary tuberculosis patients aged 18-65 years old ，each dose for10 cases.
  Interventions: Biological: Recombinant Mycobacterium Tuberculosis Fusion Protein (EEC)
- Healthy subjects (Experimental): Experimental drug of low-dose (2.5 μg/ml), medium-dose (5 μg/ml), and high-dose (10 μg/ml) will be conducted separately for 30 healthy subjects aged 18-65 years old ，each dose for10 cases.
  Interventions: Biological: Recombinant Mycobacterium Tuberculosis Fusion Protein (EEC)

INTERVENTIONS:
Biological: Recombinant Mycobacterium Tuberculosis Fusion Protein (EEC) — 1.0ml/bottle, containing 2.5μg/ml low dose, 5μg/ml medium dose, and 10μg/ml high dose of active ingredient.
  Take 0.1ml and inject it into the center of the front 1/3 of the palm side of the forearm by the Montessori method Single dose administration.

SUMMARY:
The study is to enroll 60 participants aged 18-65 years old, including 30 healthy subjects and 30 tuberculosis patients. Low-dose (2.5 μg/ml), medium-dose (5 μg/ml), and high-dose (10 μg/ml) studies will be conducted separately for healthy subjects and pulmonary tuberculosis patients, with 20 participants in each dosage group. Within 28 days after the skin test of the test drug, observations were made of reactions at the skin test site, reactions at non-skin test sites, concomitant medication, and any other physical discomfort (skin test site-specific reactions were recorded separately).

DETAILED DESCRIPTION:
The study is to enroll 60 participants aged 18-65 years old, including 30 healthy subjects and 30 tuberculosis patients. Low-dose (2.5 μg/ml), medium-dose (5 μg/ml), and high-dose (10 μg/ml) studies will be conducted separately for healthy subjects and pulmonary tuberculosis patients, with 20 participants in each dosage group.

Enrollment will progress from low to high dosages, first with healthy subjects and then with pulmonary tuberculosis patients. The safety review committee (SRC) will review safety data before each dosage group escalates and before enrollment of tuberculosis patients. See the figure below for details.

First, 10 healthy subjects will be enrolled in the low-dose group. After confirming the safety of the test drug within 72 hours of the skin test for all participants, the medium-dose group (10 participants) will be enrolled. After confirming the safety of the test drug within 72 hours of the skin test for all participants, the high-dose group (10 participants) will be enrolled. Participants will receive a single intradermal injection of 0.1 ml of the test drug using the Mantoux method on the volar aspect of the forearm.After the last healthy subject in the low-dose group completes the 72-hour safety assessment following the skin test, pulmonary tuberculosis patients in the low-dose group can be enrolled simultaneously.

Ten pulmonary tuberculosis patients will be enrolled in the low-dose group. After confirming the safety of the test drug within 72 hours of the skin test for all participants, the medium-dose group (10 participants) will be enrolled. After confirming the safety of the test drug within 72 hours of injection for all participants, the high-dose group (10 participants) will be enrolled. Participants will receive a single intradermal injection of 0.1 ml of the test drug using the Mantoux method on the volar aspect of the forearm.

Within 28 days after the skin test of the test drug, observations were made of reactions at the skin test site, reactions at non-skin test sites, concomitant medication, and any other physical discomfort (skin test site-specific reactions were recorded separately).

ELIGIBILITY:
Inclusion Criteria:

* For healthy participants：

  1. Age 18 to 65 years old (including 18 and 65), both males and females are eligible;
  2. Willing to participate in the trial and sign an informed consent form;
  3. Able to comply with the requirements of the clinical trial protocol and participate in follow-up;
  4. No history of tuberculosis (including pulmonary and extrapulmonary tuberculosis), no family history of tuberculosis (in direct relatives), and no history of close contact with tuberculosis patients (referring to direct contact with registered tuberculosis patients within 3 months before their diagnosis or within 14 days after starting anti-tuberculosis treatment);
  5. No clinical symptoms of tuberculosis poisoning; chest X-ray examination is normal or abnormal but has no clinical significance; vital signs: body temperature (axillary temperature) <37.3℃, blood pressure (systolic pressure <140mmHg, diastolic pressure <90mmHg), pulse 50~100 times/min, electrocardiogram, physical examination is normal or abnormal but has no clinical significance;
  6. Laboratory tests including blood routine, urine routine, and blood biochemistry are normal or abnormal but have no clinical significance;
  7. Female participants of childbearing age must have a negative pregnancy test before enrollment and have no plans to conceive within 28 days after enrollment, and promise to take effective contraceptive measures (including: oral contraceptives, injection or implantation of contraceptives, slow-release local contraceptives, hormonal patches, intrauterine devices (IUD), sterilization, avoidance of sexual activity, condoms (male), diaphragms, cervical caps, etc.; contraceptive methods such as safe period contraception, coitus interruptus, and emergency contraception are not considered effective).
* For patients with pulmonary tuberculosis

  1. Diagnosed as pulmonary tuberculosis according to the "Diagnostic Criteria for Pulmonary Tuberculosis in the Health Industry Standard of the People's Republic of China (WS288-2017)" (recognized clinical diagnosis made through comprehensive analysis);
  2. Aged 18 to 65 years old (including 18 and 65), regardless of gender;
  3. Willing to participate in this trial and sign an informed consent form;
  4. Able to comply with the requirements of the clinical trial protocol and participate in follow-up visits;
  5. Women of childbearing age must have a negative pregnancy test before enrollment, have no plans to conceive within 28 days after enrollment, and commit to using effective contraception (including oral contraceptives, injection or implantation of contraceptives, slow-release local contraceptives, hormone patches, intrauterine devices (IUDs), sterilization, avoiding sexual activity, male condoms, diaphragms, cervical caps, etc.; ineffective contraceptive measures include the safe period method, withdrawal method, and emergency contraception, etc.)

Exclusion Criteria:

* Known or suspected (or with a high risk of occurrence) immune dysfunction or abnormalities, including : ①Patients receiving immunosuppressive agents (including chemotherapy) or immunostimulants;②Patients who have received immunoglobulin preparations or blood products or plasma extraction treatment within the past 3 months;③Patients with malignant tumors, AIDS, etc.;
* History of seizures, epilepsy, or psychiatric illness and/or family history of psychiatric illness (first-degree relatives);
* Allergic constitution, such as a history of allergies to two or more drugs or foods, or known allergies to the components of the drug or a keloid-prone constitution;
* Currently suffering from acute infectious diseases (such as measles, pertussis, influenza, pneumonia, etc.), acute conjunctivitis, acute otitis media, or widespread skin diseases;
* Past or present history of severe cardiovascular, liver, kidney, gastrointestinal, neurological, psychiatric or metabolic abnormalities, etc., as determined by questioning;
* Acute febrile illness;
* Severe infection (such as pyoderma, severe eczema, etc.);
* Currently participating or having participated in any other new drug clinical trial within the past 3 months;
* Pregnant or lactating women;
* Drug abusers or alcoholics;
* Any other situation that the researcher believes may affect the evaluation of the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) at the skin test site and non-skin test site within 28 days after skin testing, with particular attention to the incidence of AEs within 7 days after skin testing. | 28 days after injection
Incidence of abnormal blood routine, blood biochemistry, urine routine, and electrocardiogram detection indexes on the 3rd day after skin testing. | 3 days after injection
Incidence of abnormal vital signs within 7 days after skin testing. | 7 days after injection
Incidence of serious adverse events (SAEs) within 28 days after skin testing. | 28 days after injection

SECONDARY OUTCOMES:
Specific skin reactions at the skin test site at 30 minutes, 2 hours, 4 , 8 , 24 , 48 , 72 , 96 hours, and 7 days after skin testing for different doses of EEC. | 7 days after injection
Agreement between skin test results and IGRA test results for different doses of EEC. | 7 days after injection
Agreement between IGRA test results before and after skin testing. | 7 days after injection

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No